CLINICAL TRIAL: NCT06709846
Title: Magnetic Resonance Imaging in Metabolic Diseases
Status: Recruiting | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Martin Heni, Prof. Dr. med., University of Ulm
Other Study IDs: 221/24
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-11

CONDITIONS: Metabolic Diseases
Keywords: Metabolic Diseases; Magnetic Resonance Imaging; Body Composition
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with Metabolic Diseases
- Healthy Control Participants

SUMMARY:
This study aims to leverage structural, functional, and metabolic magnetic resonance imaging (MRI) of the brain to identify imaging features that correlate with clinical parameters. It is hypothesized that individuals with metabolic diseases exhibit distinct functional and structural brain differences compared to healthy controls. These differences may evolve over time due to changes in whole-body metabolism or body weight, influenced by factors such as the natural progression of the disease or therapeutic interventions. Additionally, potential brain changes may correlate with body composition metrics, such as the fat content of specific body compartments.

This is a prospective, single-center study conducted at Ulm University Hospital, designed to track the clinical and imaging histories of patients with metabolic diseases and compare them to healthy individuals. Eligible participants include adults (aged 18 and older) capable of providing informed consent. Recruitment will occur through routine clinical care or existing research studies. To provide a comprehensive understanding, the study will include both cross-sectional analyses and longitudinal follow-up of participants, integrating repeated assessments during routine medical visits.

ELIGIBILITY:
Inclusion Criteria:

* patients with metabolic diseases OR
* healthy control participants without metabolic diseases
* written consent

Exclusion Criteria:

* History of traumatic brain injuries
* preterm birth (≤34th week of pregnancy) of the study participant
* history of brain surgery
* structural brain changes (e.g., tumors, congenital abnormalities, etc.)
* neurological developmental disorders (e.g., autism spectrum disorders, learning disabilities, intellectual disability)
* epilepsy,
* drug addiction
* other severe neurological or severe psychiatric disorders (e.g., schizophrenia
* pregnancy
* acute clinically relevant inflammatory diseases
* acute systemic or local infections
* severe or etiologically unclear diseases depending on the principle investigators judgement
* pre-existing intellectual impairment
* significant limitations in language comprehension
* absence of written consent
* general exclusion criteria for MRI imaging (e.g., pacemaker systems, neurostimulators, cochlear implants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Besides healthy controls, we will include patients who are treated for metabolic diseases at Ulm University Hospital. After the scan for cross-sectional assessment (baseline), patients who are clinically followed up at Ulm University Hospital will be offered follow-up scans, depending on changes in body weight or metabolism.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2025-02-08 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Structural differences in the brain between patients with metabolic diseases and healthy controls | cross-sectional and up to 5 years, depending on regular visits as part of routine patient care that, however, are not part of this scientific project.
  Comparison of brain anatomical magnetic resonance imaging sequences (T1- and T2-weighted sequences) between patients with metabolic diseases and healthy controls give insights into structural features in patients with metabolic diseases.
Functional differences in the brain between patients with metabolic diseases and healthy controls | cross-sectional and up to 5 years, depending on regular visits as part of routine patient care that, however, are not part of this scientific project.
  Comparison of brain functional magnetic resonance imaging between patients with metabolic diseases and healthy controls will give insights into functional aspects of patients with metabolic diseases.
Metabolic differences in the brain between patients with metabolic diseases and healthy controls | cross-sectional and up to 5 years, depending on regular visits as part of routine patient care that, however, are not part of this scientific project.
  Comparison of brain metabolic magnetic resonance imaging (Chemical Exchange Saturation Transfer (CEST)", MR-spectroscopy) between patients with metabolic diseases and healthy controls give insights into metabolic features in patients with metabolic diseases
Body Composition derived from magnetic resonance imaging | cross-sectional and up to 5 years, depending on regular visits as part of routine patient care that, however, are not part of this scientific project.
  Magnetic resonance imaging (DIXON sequence or fat-water imaging to determine the "Proton Density Fat Fraction" (PDFF)) will be used to determine the fat content in the different compartments of the whole body.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: Undecided